CLINICAL TRIAL: NCT05635877
Title: Effects of Low-dose Esmolol on Myocardial Injury After Non-cardiac Surgery in Elderly Frail Patients:A Multicenter, Prospective, Double-blind, Randomized Controlled Study
Brief Title: Effects of Low-dose Esmolol on Myocardial Injury After Non-cardiac Surgery in Elderly Frail Patients
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Yongtao Sun (Other)
Responsible Party: Sponsor-Investigator, Yongtao Sun, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20221028YTsun
Record Dates: First submitted 2022-11-03; First posted 2022-12-02 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Frailty; Esmolol; Myocardial Injury
Keywords: myocardial injury after non-cardiac surgery, MINS
MeSH Terms: conditions — Frailty | interventions — esmolol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Esmolol (Experimental): The treatment group was given esmolol 0.5mg/kg load, 10μg /kg/min continuous pump; Patient-controlled analgesia pump (sufentanil 2 μg/kg, 2 mL/h, for 48h) was used as the postoperative analgesia regimen in the two groups. If the VAS score was >3, analgesic adjuvant drugs were given intravenously and recorded. If repeated treatment is ineffective, the study will be excluded.
  Interventions: Drug: Esmolol
- Placebo Comparator:normal saline(0.9%) (Placebo Comparator): The control group received the same volume of 0.9% normal saline, which was continuously pumped until the end of the operation before extubation.Patient-controlled analgesia pump (sufentanil 2 μg/kg, 2 mL/h, for 48h) was used as the postoperative analgesia regimen in the two groups. If the VAS score was >3, analgesic adjuvant drugs were given intravenously and recorded. If repeated treatment is ineffective, the study will be excluded.
  Interventions: Drug: Placebo Comparator: Placebo Comparator:normal saline(0.9%)

INTERVENTIONS:
Drug: Esmolol — The treatment group was given Esmolol 0.5mg/kg load and 10μg /kg/min continuous pump
  Arms: Experimental:Esmolol
Drug: Placebo Comparator: Placebo Comparator:normal saline(0.9%) — The control group received the same volume of 0.9% normal saline, which was continuously pumped until the end of the operation before extubation.Patient-controlled analgesia pump (sufentanil 2 μg/kg, 2 mL/h, for 48h) was used as the postoperative analgesia regimen in the two groups. If the VAS score was >3, analgesic adjuvant drugs were given intravenously and recorded. If repeated treatment is ineffective, the study will be excluded.
  Arms: Placebo Comparator:normal saline(0.9%)

SUMMARY:
This topic will focus on the following questions:

1. Part one: To clarify the relationship between preoperative frailty and myocardial injury (cTnT ≥0.03) after non-cardiac surgery in elderly patients; To further explore the predictive factors of myocardial injury after non-cardiac surgery （MINS） in elderly frail patients before operation.
2. Part Two: To explore the effect of low-dose esmolol on myocardial injury after non-cardiac surgery in frail elderly patients.

DETAILED DESCRIPTION:
Esmol is a short-acting selective β-adrenergic receptor blocker, which is often used in patients with cardiovascular diseases or hypertension. It is also used to reduce stress response, control heart rate and reduce myocardial oxygen consumption during perioperative period to effectively protect cardiac function. However, the safety and efficacy of perioperative β-blockers are still controversial due to their possible effects on renal function. Several recent studies have shown that β-blockers reduce perioperative myocardial ischemia and may reduce the risk of perioperative myocardial infarction (PMI) and cardiovascular death in high-risk patients . The 2021 American College of Cardiology /American Heart Association (ACC/AHA )guidelines for coronary revascularization suggest that dose adjustment can optimize the clinical effects of β-blockers, thereby reducing adverse effects during treatment . In addition, several studies have found that continuous intraoperative infusion of low-dose esmolol (5-10μg/kg/min) can reduce intraoperative stress response and maintain hemodynamic stability. The meta-analysis of esmolol by Ollila A et al. found that esmolol has a promising application in the prevention of perioperative myocardial ischemia and serious complications associated with long-term ischemia. Does perioperative Esmolol reduce the incidence of myocardial injury after non-cardiac surgery （MINS）? The safety, outcome and benefit of perioperative esmolol in frail patients are still unclear. Therefore, this study intends to apply the appropriate dose of esmolol to prevent cardiovascular events in elderly frailty patients undergoing non-cardiac surgery, and explore the effect of low-dose esmolol on MINS in elderly frail patients, so as to provide feasible clinical measures for the safe outcome and rehabilitation of frail patients during perioperative period.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years;
2. ASA: ⅰ-ⅳ;
3. Modified frailty index (mFI) ≥ 0.21;
4. Patients undergoing non-cardiac surgery.

Exclusion Criteria:

1. Refuse to participate;
2. Expected hospital stay <3 days;
3. Preoperative β-blocker therapy;
4. History of myocardial infarction or coronary artery disease;
5. Preoperative bradycardia (heart rate [HR] < 50 bpm) or arrhythmia;
6. Significant cardiac insufficiency (i.e., pulmonary artery pressure >18 mm Hg, cardiac index ≤ 2.2 L/min/m 2);
7. Severe valvular heart disease;
8. Severe lung disease (e.g. asthma or chronic obstructive pulmonary disease);
9. Patients with perioperative troponin elevation due to nonischemic causes (e.g., sepsis, pulmonary embolism, arrhythmia);
10. The same patient can only be included once, regardless of whether the reason for the second operation is related to the first cause.

    -

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2023-02-07 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
incidence of Postoperative myocardial injury after non-cardiac surgery(MINS) | incidence of MINS within 3 days after operation
  incidence of Postoperative myocardial injury after non-cardiac surgery（MINS）, blood samples were collected at 1 day before surgery and 1, 2, and 3 days after surgery.
  MINS diagnostic criteria: Blood samples were collected before surgery, 1d, 2d and 3d after surgery for Roche fourth-generation Elecsys hs-TnT detection, cardiac troponin（cTnT） ≥ 0.03 ng/mL, and MINS can be diagnosed.

SECONDARY OUTCOMES:
the results of 30 days after surgery | Outcomes at 30 days after operation were recorded
  the results of 30 days after surge, demographic characteristics of patients, preoperative disease complications, the treatments number of intraoperative hemodynamic instability , hospital stays, any complications occurring within 30 days after surgery, and readmitted to hospital were recorded.
  Perioperative MAP < 65 mmHg or bradycardia (HR) < 50 times /min in both groups, and no spontaneous remission was found 5 minutes after the operation was stopped, that is, intervention measures were given, including ephedrine, atropine, dopamine and other treatments., demographic characteristics of patients, preoperative disease complications, the number of intraoperative hemodynamic instability treatments, length of stay, any complications occurring within 30 days after surgery, and readmitted to hospital were recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Derived] Sun Y, Guo N, Zhang M, Liu M, Gao Z, Sun T, Gao X, Xu L, Zhang H, Wei C, Liu P, Liu Y, Zhang X, Guo Y, Chen L, Zhou Z, Su Z, Hu Y, Shi X, Huang L, Wang Y. Association between preoperative frailty and myocardial injury after noncardiac surgery in geriatric patients: study protocol for a prospective, multicentre, real-world observational, cohort trial. BMC Geriatr. 2024 Mar 19;24(1):271. doi: 10.1186/s12877-024-04847-z. PMID 38504166